CLINICAL TRIAL: NCT05753566
Title: Efficacy and Safety of Rezvilutamide in Patients With Biochemical Recurrence After Radical Prostatectomy for Prostate Cancer: A Prospective, Multi-centre Study
Brief Title: Rezvilutamide in Patients With Biochemical Recurrence After Radical Prostatectomy for Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hongqian Guo, Chief physician of Department of Urology, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-119
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer; Biochemical Recurrence
Keywords: Prostate cancer; Biochemical recurrence; Rezvilutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rezvilutamide +ADT+ SRT (Experimental): Rezvilutamide along with ADT for 6 cycles (28 days for each cycle) in combination with salvage radiation therapy (SRT) according to standard of care
  Interventions: Drug: Rezvilutamide; Drug: Androgen deprivation therapy (ADT); Radiation: SRT
- Rezvilutamide +ADT (Experimental): Rezvilutamide along with ADT for 12 cycles (28 days for each cycle)
  Interventions: Drug: Rezvilutamide; Drug: Androgen deprivation therapy (ADT)

INTERVENTIONS:
Drug: Rezvilutamide — Specifications of 80 mg; orally, once a day
  Other Names: SHR3680
Drug: Androgen deprivation therapy (ADT) — Androgen deprivation therapy (ADT), the ADT used by each subject will be determined by the investigator, and the dose and frequency of administration will be consistent with the prescription information
Radiation: SRT — SRT according to standard of care (66.6-72 grays will be delivered to the bed of prostate ,~50.4 grays to the pelvis if needed)
  Arms: Rezvilutamide +ADT+ SRT

SUMMARY:
To evaluate the efficacy and safety of rezvilutamide in combination with androgen deprivation therapy(ADT) and standard salvage radiation therapy(SRT) or rezvilutamide in combination with ADT in prostate cancer patients with biochemical recurrence of prostate-specific antigen(PSA) persistence after radical prostatectomy(RP).

ELIGIBILITY:
Main Inclusion Criteria:

1. Age ≥ 40 years, male.
2. Patients with histologically-confirmed diagnosis of prostate adenocarcinoma.
3. pathologically node-negative (pN0) or pathologically node cannot be assessed (pNx);
4. Patients with PSA < 0.1ng/ml within 8 weeks after radical prostatectomy (RP) and maintained for at least 6 months;
5. Biochemical recurrence (two consecutive rises in PSA with absolute values > 0.2ng/ml, the time interval ≥ 2 weeks apart ) and no local recurrence or distant metastatic lesions on conventional imaging (bone scan and CT/MRI scan);
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1;
7. Estimated life expectancy >10 year;
8. Adequate laboratory parameters

   * Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9/L
   * Platelet count (PLT) ≥ 100 x 10^9/L
   * Haemoglobin (Hb) ≥ 90 g/L
   * Serum creatinine (Cr) ≤ 1.5 x upper limit of normal(ULN) or creatinine clearance > 50 ml/min.
   * Total bilirubin (TBIL) ≤ 1.5 x ULN.
   * Glutamic oxaloacetic transaminase (AST/SGOT) or glutamic alanine transaminase (ALT/SGPT) levels ≤ 2.5 x ULN.
   * International normalised ratio (INR) ≤1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT)≤1.5 x ULN .
   * Left ventricular ejection fraction (LVEF) ≥ 50%.
9. Patients able to comply with the protocol. Arm 1 subjects are proposed to receive salvage radiation therapy, while arm 2 subjects are not suitable for or refuse radiation therapy.
10. Signed informed consent.

Main Exclusion Criteria:

1. Prior hormonal therapy (antiandrogens or gonadotropin releasing hormone) or prior radiotherapy to pelvic .
2. Postoperative biochemical recurrence with PSA > 2 ng/ml.
3. Postoperative pathology containing neuro-endocrine differentiation or small cell features.
4. Prior malignancy other than prostate cancer in the past three years.
5. History of any of the following:

   * Seizure or known condition that may pre-dispose to seizure
   * Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to entry.
   * Active infection (eg, human immunodeficiency virus [HIV] or viral hepatitis)
6. Any other serious or uncontrolled illness which in the opinion of the investigator makes it undesirable for the patient to enter the trial.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
2-year biochemical progression-free survival | 24 months
  For arm 1, biochemical progression is defined as a confirmed prostate specific antigen (PSA) greater than (>) 0.2 nanogram per milliliter (ng/ml)
3-year biochemical progression-free survival | 36 months
  For arm 2, biochemical progression is defined as a confirmed PSA greater than (>) 0.2 ng/ml( the time interval should be over 2 weeks)

SECONDARY OUTCOMES:
biochemical progression-free survival | 36 months
  Time from entry to biochemical progression or death due to any cause.
progression-free survival (PFS) | 36 months
  Time from entry to biochemical progression or radiologically confirmed progressive disease or death due to any cause.
metastasis-free survival (MFS) | 36 months
  Time from entry to radiologically confirmed metastasis disease or death due to any cause.
Quality of life as determined by FACT-P scores | At baseline, 3 months, 6 months, every 3 months up to 3 years
  Quality of life as determined by Functional Assessment of Cancer Therapy-Prostate (FACT-P) scores
Quality of life as determined by EPIC-26 questionnaire | At baseline, 3 months, 6 months, every 3 months up to 3 years
  Quality of life as determined by Expanded Prostate Cancer Index Composite-26 (EPIC-26) questionnaire
Number of Adverse Events | 36 months
  Number of Adverse Events
Duration of testosterone recovery | 36 months
  Duration of testosterone recovery
Time to testosterone recovery to >50 ng/dl | 36 months
  Time to testosterone recovery to >50 ng/dl
Time to testosterone recovery to >300 ng/dl | 36 months
  Time to testosterone recovery to >300 ng/dl

CONTACTS AND LOCATIONS:
Overall Officials: Chief physician of Department of Urology, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (2):
- China (2):
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - JiangSu Cancer Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No